CLINICAL TRIAL: NCT00287365
Title: Glutathione S Transferase M1 (GSTM1) Genotype Associated Susceptibility to Airway Response to Ozone in Mild Asthmatic Volunteers.
Brief Title: Genetic Susceptibility to Ozone in Mild Asthmatic Volunteers
Acronym: Glutoz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GCRC-2371; NCCAM 1PO1AT002620 (Other Grant/Funding Number: National Center for Complementary and Alternative Medicine)
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Mild Asthma
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1-ozone (Experimental): Mildly asthmatic subjects with GSTM1 null genotype compared to GSTM1 sufficient subjects
  Interventions: Drug: ozone

INTERVENTIONS:
Drug: ozone — 2 hour exposure to 0.4 ppm ozone
  Other Names: O3

SUMMARY:
Recent reports have shown that people with asthma who have a particular gene, known as the GSTM1 null gene, are more susceptible to the effect of air pollutants. The purpose of this research study is to learn if volunteers who have asthma and have a GSTM1 null gene have increased response (change in lung function and increase in lung cells collected from sputum) compared to volunteers with asthma who have the GSTM1 sufficient gene when challenged with 0.4 ppm ozone during intermittent exercise. The principal purpose of this study is to identify hyper-responsive, responsive and non-responsive groups of human subjects with mild asthma based on their airway neutrophilic response to ozone exposure, and to perform analyses on DNA from airway cells to explore possible differences in genetic profiles between the three groups. An additional pilot aim is to compare expression of a small number of specific genes of interest in a subset of ozone-responsive and ozone-non-responsive subjects with mild asthma.

DETAILED DESCRIPTION:
Fifty volunteers with mild asthma will be recruited to undergo ozone challenge in the controlled exposure facility of the US EPA Human Studies Division (104 Mason Farm Road, Chapel Hill, NC) with 0.4ppm for 2 hours with moderate exercise alternating with rest. Endpoints will include genetic analysis for the GSTM1 genotype, sputum and spirometry changes pre and post exposure, and blood endpoints pre and post exposure.

TRAINING DAY: (at least 3 days prior to the ozone challenge) Eligible subjects will report to the research lab for a 3 hour training session.

* All female volunteers will undergo a urine pregnancy test.
* After informed consent is obtained, Measurement of orally exhaled nitric oxide will be obtained
* Subjects will perform spirometry.
* Subjects will exercise on a treadmill to determine the workload for the actual exposure.
* Finally the subject will undergo sputum induction following pretreatment with albuterol.

The sputum will be assessed for quality to determine continued eligibility. If a subject has provided an acceptable sputum sample within the prior 6 months this may be used as inclusion criteria rather than repeating the induction at this point. After subjects have demonstrated production of an adequate sputum sample, they will be scheduled for the ozone exposure visit.

24 HOURS PRIOR to the exposure day (Day 1): Subjects will be asked to refrain from smoking as well as drinking alcohol for 24 hours prior to Day 1 until after completion of Day 3.

* Subjects will have vital signs and oxygen saturation checked, including the symptom questionnaire.
* They will also undergo a physical examination of the ears, nose, throat and chest (lung sounds).
* Female volunteers will undergo urine pregnancy testing.
* Measurement of orally exhaled nitric oxide will be obtained.
* Spirometry testing will be performed.
* Subjects will have a sputum induction preceded by administration of 2 puffs of albuterol.

EXPOSURE DAY (at least 3 days after the training day):

* Subjects will be asked to arrive at the study site at approximately 8 AM and will undergo assessment of vital signs (temperature, pulse, respiratory rate, blood pressure), oxygen saturation, and symptom score assessment.
* A telemetry unit will be placed for cardiac monitoring during the exposure.
* Measurement of orally exhaled nitric oxide will be obtained prior to exposure and 4 hours after the end of the exposure
* Spirometry testing to rule out acute illness prior to the exposure.
* They will also undergo a physical examination of the ears, nose, throat and chest.
* Exposure sessions: The 0.4 ppm ozone exposure will be conducted in an ozone exposure chamber. Each subject will be exposed to 0.4 ppm ozone for 2 hours. During exposures, subjects will perform four 15 minute bouts of moderate exercise (minute ventilation or VE = 30 40 L/min) on a treadmill, each separated by 15 minutes of seated rest. Minute ventilation is measured for 2 to 3 minutes after about 4 minutes of exercise during the first exercise period, and again at about 12 minutes of exercise. It is then measured at about 12 minutes into each exercise period. Two subjects may be exposed simultaneously, in which case the exercise/rest periods will be alternated.
* Immediately post exposure and 4 hours after completion of exposure, subjects will have an assessment of vital signs, oxygen saturation, symptom score assessment and undergo spirometry evaluation.
* Venipuncture: 20 ml of blood will be collected for a CBC/ differential, assessment of blood monocyte phagocytic function and cell surface markers just prior to the exposure and 4 hours after the end of exposure. A portion of the sample will be used for genotyping.
* Induced sputum will be collected 6 hours after initiation of exposure after subjects have been premedicated with albuterol. The subjects will be observed at the study site until sputum induction is complete. Subjects will not be discharged home following the post-exposure sputum induction until FEV1 is within 90% of baseline values and vital signs are normal. Subjects not meeting safety criteria at the end of the exposure day will be admitted to the GCRC for overnight observation.

  24 HOURS POST EXPOSURE (Day 3): The following morning, approximately 24 hours after exposure, the volunteer subject will be assessed directly at the study site. The subject will undergo spirometry, vital sign monitoring and symptom scoring.

STUDY DISCONTINUATION VISIT (5-10 days after exposure): The volunteer subject will again be assessed directly at the study site. The subject will undergo spirometry, vital sign monitoring and symptom scoring.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with mild asthma
* Normal lung function,
* Oxygen saturation of > 94 %
* Normal blood pressure

Exclusion Criteria:

* A history of significant chronic illnesses
* Allergy to any medications which may be used or prescribed in the course of this study (albuterol, acetaminophen, aspirin or non-steroidal anti-inflammatory agents, corticosteroids, lactose, polyethylene glycol)
* Positive pregnancy test within 48 hours of the time of challenge
* Subjects currently taking medications which may impact the results of the ozone challenge, interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents) or suggest an ongoing illness (such as antibiotics).
* Mega doses of vitamins and supplements, homeopathic/naturopathic medicines
* Any acute, non-chronic, medical conditions occurring in the prior two weeks. Such illnesses must be totally resolved symptomatically for 2 weeks and documentation of normal lung function must be obtained.
* Unspecified illnesses, which in the judgment of the investigator might increase the risk associated with ozone inhalation challenge, will be a basis for exclusion.
* Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
* Use of systemic steroid therapy within the preceding 12 months.
* > 0.5 pack year history of tobacco use
* Use of inhaled steroids, cromolyn or leukotriene inhibitors initiated within the past month (except for use of cromolyn exclusively prior to exercise). Patients must be on a stable regimen of therapy.
* Use of daily theophylline within the past month.
* Pregnancy or nursing a baby.
* Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Exacerbation of asthma more than 2x/week which would be characteristic of a person with moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
* Dosing level of an inhaled steroid must be consistent with mild episodic asthma as outlined by the NHLBI NAEPP guidelines. Use of inhaled steroid at doses typically used for moderate or severe asthma will result in exclusion of that individual from the protocol.
* Students or staff members who work directly for the PI, Dr David Peden, are excluded from study participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B. Peden, MD, Principal Investigator — University of NC Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Center for Environmental Medicine, Asthma and Lung Biology — http://www.med.unc.edu/cemalb/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: None. All subjects who successfully screened were enrolled.
Groups:
- Mildly Asthmatic Subjects With GSTM1 Null Genotype Compared to: Mildly asthmatic subjects with GSTM1 null genotype compared to GSTM1 sufficient subjects
  ozone: 2 hour exposure to 0.4 ppm ozone
Period: Overall Study
Arm/Group | Mildly Asthmatic Subjects With GSTM1 Null Genotype Compared to
Started | 25
Completed | 12
Not Completed | 13
Not completed — sample not acquired | 13

BASELINE CHARACTERISTICS:
Population: Analysis population only includes those who could produce sputum after ozone challenge. 2 of the original 25 volunteers did not produce adequate sputum
Arm/Group | Mildly Asthmatic Subjects With GSTM1 Null Genotype Compared to
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 25 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 subjects had insufficient sputum post exposure for analysis.
  Participants
    Female | 8
    Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Post Ozone Change in Lung Function (FEV1) Between Subjects With GSTM1 Null Genotype Compared to GSTM1 Sufficient Subjects
Time Frame: 6 hours post exposure
Population: Mild asthmatics exposed to ozone
Measure: Mean (Standard Error); unit: percentage of FEV1 predicted
Groups:
- GSTM1 Null: GSTM1 null mild asthmatics
- GSTM1 Sufficient: GSTM1 sufficient mild asthmatics
Arm/Group | GSTM1 Null | GSTM1 Sufficient
Number analyzed (Participants) | 4 | 8
percentage of FEV1 predicted | 85 (6) | 79 (6)

2. Secondary Outcome: Secondary Endpoints Include Post Ozone Airway PMN Influx Between Subjects With GSTM1 Null Genotype Compared to GSTM1 Sufficient Subjects
Time Frame: 6 hours post exposure
Measure: Mean (Standard Error); unit: percentage of cells
Arm/Group | GSTM1 Null | GSTM1 Sufficient
Number analyzed (Participants) | 4 | 8
percentage of cells | 4 (8) | 8 (16)

3. Secondary Outcome: % Decrease in FVC in Asthmatics Between Subjects With GSTM1 Null Genotype Compared to GSTM1 Sufficient Subjects
Time Frame: 6 hours post exposure
Measure: Mean (Standard Error); unit: percentage of FVC predicted
Arm/Group | GSTM1 Null | GSTM1 Sufficient
Number analyzed (Participants) | 4 | 8
percentage of FVC predicted | 93 (5) | 85 (4)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Mildly Asthmatic Subjects With GSTM1 Null Genotype Compared to
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mildly Asthmatic Subjects With GSTM1 Null Genotype Compared to (N=25)
decreased FEV1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No